CLINICAL TRIAL: NCT05369910
Title: How Can we Treat Photophobia in Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Austrian Science Fund (FWF) (Other)
Responsible Party: Principal Investigator, Dr. Eva Matt, Research assistant, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KLI 455
Record Dates: First submitted 2022-05-02; First posted 2022-05-11 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Migraine Disorders; Photophobia
Keywords: migraine; photophobia; habituation; headache; functional magnetic resonance imaging
MeSH Terms: conditions — Migraine Disorders; Photophobia; Substance-Related Disorders; Headache

STUDY DESIGN:
Intervention Model Description: Participants receive light exposure therapy (Flash) and light deprivation therapy (Dark) for one hour daily on 7 consecutive days, in a crossover design with a wash-out period of 3 months. The sequence of the interventions is randomly allocated.
Masking Description: Due to the nature of the interventions, no blinding is possible, but both Flash and Dark interventions are presented as equivalently treatment options.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flash first (Experimental): Light exposure (Flash) first, light deprivation (Dark) second:
  Both interventions (Flash and Dark) are administered for one hour on 7 consecutive days. During the light exposure, participants are seated 120 cm in front of a white curtain that is illuminated by an LED light source. During the light deprivation, participants are seated in the same room used for light exposure, but in complete darkness.
  Interventions: Behavioral: Light exposure (Flash); Behavioral: Light deprivation (Dark)
- Dark first (Experimental): Light deprivation (Dark) first, Light exposure (Flash) second:
  Both interventions (Flash and Dark) are administered for one hour on 7 consecutive days. During the light exposure, participants are seated 120 cm in front of a white curtain that is illuminated by an LED light source. During the light deprivation, participants are seated in the same room used for light exposure, but in complete darkness.
  Interventions: Behavioral: Light exposure (Flash); Behavioral: Light deprivation (Dark)

INTERVENTIONS:
Behavioral: Light exposure (Flash) — Light exposure (Flash) is administered for one hour on 7 consecutive days. During the light exposure, participants are seated 120 cm in front of a white curtain that is illuminated by an LED light source (Dawe stroboscope type 1214B, 5 Hz).
Behavioral: Light deprivation (Dark) — Light deprivation (Dark) is administered for one hour on 7 consecutive days. During the Dark intervention, participants are seated in a room in complete darkness.

SUMMARY:
Photophobia, the aberrantly increased sensitivity to light, is a common symptom in migraine patients and light discomfort is frequently found as a trigger for migraine attacks. In behavioral studies, planned exposure to light was found to reduce headache in migraineurs with photophobia, potentially by increasing habituation to this migraine trigger. Here, neurophysiological mechanisms of light exposure versus light deprivation therapy in migraine patients are investigated using functional magnetic resonance imaging (fMRI).

Migraine patients and healthy controls receive light exposure therapy (Flash) and light deprivation therapy (Dark) for one hour daily on 7 consecutive days, in a crossover design with a wash-out period of three months. Study participants keep a diary including items on interictal and ictal photophobia, headache frequency and severity 7 days before, during, and 7 days after the interventions. One week before and one day after both interventions, fMRI using flickering light in a block design is applied. Functional activation is analyzed at whole-brain level and habituation of the visual cortex (V1) is modeled with the initial amplitude estimate and the corrected habituation slope.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Migraine without aura according to the criteria of the International Classification of Headache Disorders (ICHD-3 beta)
* 1-4 days with migraine per month in the preceding last 3 months
* A score between 2 and 6 on a numeric rating scale for the intensity of interictal photophobia (range from 0 to 10 (= max. intensity))
* A score >4 for ictal photophobia

Controls

* No personal or family history of migraine
* A score <2 for photophobia

Exclusion Criteria:

* Current or previous circadian rhythm disorders
* Current or previous major depression
* Current or previous anxiety disorders
* Current or previous medication overuse
* Besides migraine in the patient group, participants should not suffer from any other recurrent headache apart from infrequent tension-type headaches

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline interictal photophobia during and after the interventions | Change in interictal photophobia during the interventions (Flash and Dark, average over 7 days) and after the interventions (Post Flash, Post Dark, average over 7 days) relative to the baseline (average over 7 days before the first intervention starts).
  Subjective sensitivity to light between migraine attacks is assessed using a numeric rating scale with the range from 0 (= no photophobia) to 10 (= max. photophobia). The numeric rating scale is daily completed by the participants over the study course using a structured diary. Daily reports are averaged for the duration of the baseline phase (7 days before the first intervention starts), for the duration of the interventions (Flash and Dark, 7 days each), and for 7 days after the interventions (Post Flash, Post Dark).

SECONDARY OUTCOMES:
Change from baseline headache frequency during and after the interventions | Change in headache frequency during the interventions (Flash and Dark, average over 7 days) and after the interventions (Post Flash, Post Dark, average over 7 days) relative to the baseline (average over 7 days before the first intervention starts).
  In the structured diary, the participants report if a headache is present (1) or absent (0). Daily reports are averaged for the duration of the baseline phase (7 days before the first intervention starts), for the duration of the interventions (Flash and Dark, 7 days each), and for 7 days after the interventions (Post Flash, Post Dark).
Change from baseline headache severity during and after the interventions | Change in headache severity during the interventions (Flash and Dark, average over 7 days) and after the interventions (Post Flash, Post Dark, average over 7 days) relative to the baseline (average over 7 days before the first intervention starts).
  If a headache is present that day, questions regarding headache severity (mild (1), moderate (2), severe (3)) are completed in the structured diary. Daily reports are averaged for the duration of the baseline phase (7 days before the first intervention starts), for the duration of the interventions (Flash and Dark, 7 days each), and for 7 days after the interventions (Post Flash, Post Dark).
Change from baseline ictal photophobia during and after the interventions | Change in ictal photophobia during the interventions (Flash and Dark, average over 7 days) and after the interventions (Post Flash, Post Dark, average over 7 days) relative to the baseline (average over 7 days before the first intervention starts).
  If a headache is present that day, photophobia during the headache is assessed on a numeric rating scale with the range from 0 (= no photophobia) to 10 (= max. photophobia). Daily reports are averaged for the duration of the baseline phase (7 days before the first intervention starts), for the duration of the interventions (Flash and Dark, 7 days each), and for 7 days after the interventions (Post Flash, Post Dark).

OTHER OUTCOMES:
Change from baseline functional activation in the primary visual cortex after the interventions | fMRI one day after the completion of each intervention (Flash, Dark) is compared the the baseline fMRI measured 7 days before the first intervention starts.
  3 Tesla functional Magnetic Resonance Imaging (fMRI) is used to analyze brain activation induced by flickering light (10 functional runs, block design with 7 alternating blocks (20 s each) of flashing light (8 Hz) and darkness (140 s per run)).

CONTACTS AND LOCATIONS:
Overall Officials: Roland Beisteiner, MD, Principal Investigator — Department of Neurology, Medical University of Vienna

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Matt E, Aslan T, Amini A, Saricicek K, Seidel S, Martin P, Wober C, Beisteiner R. Avoid or seek light - a randomized crossover fMRI study investigating opposing treatment strategies for photophobia in migraine. J Headache Pain. 2022 Aug 11;23(1):99. doi: 10.1186/s10194-022-01466-0. PMID 35948966